CLINICAL TRIAL: NCT00414830
Title: Systematic Prevention of Further Fractures in Patients With Hip Fractures and Osteoporosis.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: National Board of Health, Denmark (Other Government); University of Southern Denmark (Other); Merck Sharp & Dohme LLC (Industry)
Other Study IDs: 023
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-04

CONDITIONS: Hip Fracture; Osteoporosis
Keywords: prevention; health technology assessment; population based; fracture
MeSH Terms: conditions — Hip Fractures; Osteoporosis; Fractures, Bone

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine if prevention of further fractures is possible through systematic evaluation for osteoporosis in patients with recent hip fracture

DETAILED DESCRIPTION:
Osteoporosis is a common disease characterized by an increased risk of fracture. Furthermore recent studies has revealed that patients with fractures have increased risk of renewed fracture. Most fractures in the elderly are partly attributable to osteoporosis. The most severe of these shown to be the hip fracture (HFx) which increase mortality and decrease health related quality of life and has major impact on the level of national health service. Solid evidence is available showing several interventions to reduce the risk of osteoporotic fractures. In spite of this only few HFx patients are offered examination or treatment for osteoporosis and very rare this happens on a routine basis.

In the county of Funen and Ribe in Denmark the departments of Endocrinology and Orthopedic Surgery at Odense University Hospital and Hospital of South Western Jutland therefore initiated a fracture discharge program as part of a health technology assessment (HTA) study offering evaluation for osteoporosis to HFx patients. Evaluation consists of Duel Energy X-ray Absorptiometry, Instant Vertebral Assessment, a biochemical panel, and clinical assessment followed by specific anti-osteoporotic treatment as appropriate.

The HTA study is designed as a longitudinal cohort study of patients admitted to the participating departments with a low energy HFx. Inclusion started January first 2005 and ends December 31. 2006. After the last inclusion the follow up of the last patient are set to 2 years. In the study period data will be collected on subsequent fractures, epidemiological and demographic factors, questionnaires on quality of life, and register data on mortality, use of medication, and use of health services. The control group consists of patients admitted to any other hospital in the two participating counties who are not given this systematic evaluation for osteoporosis on a routine basis.

The HTA report will provide data to suggest if a systematic offer of evaluation and treatment of osteoporosis in HFx patients:

can reduce further fractures is accepted by the majority of patients can increase the amount of life years by decreasing mortality can increase quality of life by reducing the amount of fractures is cost effective for the health care providers

ELIGIBILITY:
Inclusion Criteria:

* admitted to the department of orthopedic surgery at Odense University Hospital or Hospital of South Western Jutland with a low energy hip fracture

Exclusion Criteria:

* dementia
* pathological fracture
* severe comorbidity
* not wanting to participate

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2005-01; Study Completion 2009-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kim T Brixen, M.D.,PH.D., Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Department og Endocrinology, Odense, Denmark